CLINICAL TRIAL: NCT01678716
Title: 1) Impact Evaluation of Behavior Change Communication and Micronutrient Supplementation Interventions on Infant and Young Child Feeding (IYCF) Practices and on Childhood Stunting and Anaemia 2) Evaluation of the Public Health Impact of a Market-based Approach to Improving Diet Quality of Infants and Young Children Through the Use of Sprinkles in Bangladesh
Brief Title: Impact of Behavior Change Communications and Market-based Approach to Delivering Micronutrient Powders on Stunting, Infant Feeding Practices and Anemia in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AED ARTS/IFPRI-S-01; IFPRI-107033 (Other Grant/Funding Number: Global Alliance for Improved Nutrition)
Record Dates: First submitted 2012-08-29; First posted 2012-09-05 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Child Malnutrition; Breastfeeding; Complementary Feeding; Childhood Anemia
Keywords: Anemia; Breastfeeding; Complementary feeding; Stunting; Wasting; Underweight; Micronutrient powder; Behavior change counseling; Frontline health worker
MeSH Terms: conditions — Child Nutrition Disorders; Breast Feeding; Anemia; Growth Disorders; Cachexia; Thinness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Essential Health Care (EHC) only (Active Comparator): This arm is the basic comparison arm, which will receive the standard package of health services offered through BRAC's essential health care (basic antenatal care, basic counseling on health and nutrition through health worker home visits. In addition, a nationwide mass media campaign on IYCF practices will ensure exposure to some messages about IYCF behaviors in this arm.
  Interventions: Behavioral: Mass media
- EHC + Micronutrient Powders (Experimental): This arm will be based on the EHC platform but will also include EHC platform health workers promoting and selling the micronutrient powders.
  Interventions: Dietary Supplement: Micronutrient powders; Behavioral: Mass media
- EHC + BCC (Experimental): This arm will have a behavior chance communications intervention to improve infant and young child feeding practices. The intervention will be delivered primarily by the frontline health workers who will visit mothers in their homes and counsel them on essential IYCF practices.
  Interventions: Behavioral: EHC + BCC; Behavioral: Mass media
- EHC + BCC + Micronutrient powders (Experimental): This arm will contain both the behavior change communication and the micronutrient powder sales intervention.
  Interventions: Behavioral: EHC + BCC; Dietary Supplement: Micronutrient powders; Behavioral: Mass media

INTERVENTIONS:
Behavioral: EHC + BCC — This arm includes home visits to mothers with infants and young children. Frontline health workers will counsel and support mothers in relation to breastfeeding and complementary feeding practices
  Arms: EHC + BCC; EHC + BCC + Micronutrient powders
Dietary Supplement: Micronutrient powders — In this intervention arm, frontline health workers will visit households and promote and sell micronutrient powders to them. The micronutrient powder is sold by the brand name "Pushtikona" in Bangladesh and contains 15 micronutrients including iron, zinc, vitamin A, vitamin C, and others.
  Arms: EHC + BCC + Micronutrient powders; EHC + Micronutrient Powders
Behavioral: Mass media — A nationwide mass media campaign of TV and radio spots on infant and young child feeding practices will be aired in 2011, 2012 and 2013. All intervention arms will be exposed to this campaign.

SUMMARY:
This complex evaluation of a large-scale program uses a cluster-randomized design where 20 geographic clusters (subdistricts) were randomized to study two sets of interventions. For the evaluation of behavior change interventions only, the 20 clusters were randomized to 10 intensive and 10 non-intensive interventions areas. For a sub-study to evaluate a market-based model for delivering micronutrient powders (MNP) along with behavior change interventions, there was subsequent randomization to comparison area, MNP-only area, Behavior Change Communication (BCC)-only area and MNP+BCC areas.

DETAILED DESCRIPTION:
The design uses a repeated cross-sectional design, with multiple age-group samples for multiple outcomes [since each set of outcomes can only be assessed in the relevant age group for the outcome; e.g., exclusive breastfeeding is only assessed in children 0-6 months of age]. These include:

1. For the evaluation of behavior change intervention only:

   * 0-6 months for breastfeeding outcomes
   * 6-23.9 months for complementary feeding outcomes (in the behavior change intervention evaluation)
   * 24-48 months for child anthropometric outcomes (related to the behavior change interventions).
2. for the substudy on behavior change and micronutrient powder interventions combined - 6-23.9 months for anemia and anthropometric outcomes

A community-based random sample of children 0-6 months, 6-23.9 months, 24-48 months old was surveyed at baseline (April-June 2010). The original anemia sub-study design had proposed surveying children 6.23.9 months of age for the MNP intervention in April-June 2013 and for the behavior change intervention in April-June 2014. Based on program implementation timelines, the endline survey dates were extended by one year such that the above age groups were then sampled and surveyed in community-based surveys in April-June 2014.

Infant feeding practices will be assessed using before-after intervention-comparison area group differences between 2010, and 2013 and 2014. Specifically, breast feeding will be assessed in children 0-6 months of age (sampled separately) and complementary feeding will be assessed in children 6-23.9 months of age (sampled separately).

Stunting will be assessed in the sample of children 24-48 months of age using before-after intervention-comparison group differences between 2010 and 2014.

In addition, the investigators will evaluate the processes through which the programs roll out using a mix of qualitative and quantitative research methods. Qualitative research methods will help to understand drivers of promotion and sales of MNPs by frontline health workers, as well as household level determinants and dynamics related to enabling purchase and use of the MNP and adhering to behavioral recommendations. Quantitative surveys of frontline health workers will help document their awareness about IYCF, MNPs, training, and sales, while quantitative surveys of the households will help document household level awareness, purchase and use of MNPs and awareness and adherence to IYCF practices for children in the target age range.

ELIGIBILITY:
Inclusion Criteria:

* Child age < 60 months

Max Age: 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8800 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding (EBF) among children 0-6 months of age | 4 years after baseline
  EBF is among the eight WHO-recommended core indicators for infant and young child feeding and will be measured using recall-based survey measures
Child anthropometry (height, weight) among children 24-48 months of age | 4 years after baseline
  Child height and weight will be measured among the repeated cross-sectional of children living in the study villages. These will be converted into z-scores based on the WHO growth reference standards.
Complementary feeding among children 6-23.9 months of age | 4 years after baseline
  Complementary feeding indicators that include timely introduction of complementary feeding (infants 6-8 months), dietary diversity, minimum dietary diversity, minimum dietary diversity, are among the eight WHO-recommended core indicators for infant and young child feeding and will be measured using recall-based survey measures in this age group.
Anemia among children 6-23.9 months | 4 years after baseline
  Anemia will be measured using Hemocue

SECONDARY OUTCOMES:
Iron deficiency | 3 years
  Iron deficiency is measured using serum ferritin and serum tranferrin receptor. Assessments are done using capillary blood.

CONTACTS AND LOCATIONS:
Overall Officials: Purnima Menon, PhD, Principal Investigator — International Food Policy Research Institute; Rahul Rawat, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- International Food Policy Research Institute, Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Derived] Kim SS, Nguyen PH, Tran LM, Alayon S, Menon P, Frongillo EA. Different Combinations of Behavior Change Interventions and Frequencies of Interpersonal Contacts Are Associated with Infant and Young Child Feeding Practices in Bangladesh, Ethiopia, and Vietnam. Curr Dev Nutr. 2019 Dec 9;4(2):nzz140. doi: 10.1093/cdn/nzz140. eCollection 2020 Feb. PMID 31976385
- [Derived] Warren AM, Frongillo EA, Nguyen PH, Menon P. Nutrition Intervention Using Behavioral Change Communication without Additional Material Inputs Increased Expenditures on Key Food Groups in Bangladesh. J Nutr. 2020 May 1;150(5):1284-1290. doi: 10.1093/jn/nxz339. PMID 31943055
- [Derived] Nguyen PH, Kim SS, Tran LM, Menon P, Frongillo EA. Intervention Design Elements Are Associated with Frontline Health Workers' Performance to Deliver Infant and Young Child Nutrition Services in Bangladesh and Vietnam. Curr Dev Nutr. 2019 Jul 10;3(8):nzz070. doi: 10.1093/cdn/nzz070. eCollection 2019 Aug. PMID 31346584
- [Derived] Frongillo EA, Nguyen PH, Saha KK, Sanghvi T, Afsana K, Haque R, Baker J, Ruel MT, Rawat R, Menon P. Large-Scale Behavior-Change Initiative for Infant and Young Child Feeding Advanced Language and Motor Development in a Cluster-Randomized Program Evaluation in Bangladesh. J Nutr. 2017 Feb;147(2):256-263. doi: 10.3945/jn.116.240861. Epub 2016 Dec 28. PMID 28031374
- [Derived] Menon P, Nguyen PH, Saha KK, Khaled A, Kennedy A, Tran LM, Sanghvi T, Hajeebhoy N, Baker J, Alayon S, Afsana K, Haque R, Frongillo EA, Ruel MT, Rawat R. Impacts on Breastfeeding Practices of At-Scale Strategies That Combine Intensive Interpersonal Counseling, Mass Media, and Community Mobilization: Results of Cluster-Randomized Program Evaluations in Bangladesh and Viet Nam. PLoS Med. 2016 Oct 25;13(10):e1002159. doi: 10.1371/journal.pmed.1002159. eCollection 2016 Oct. PMID 27780198
- [Derived] Menon P, Nguyen PH, Saha KK, Khaled A, Sanghvi T, Baker J, Afsana K, Haque R, Frongillo EA, Ruel MT, Rawat R. Combining Intensive Counseling by Frontline Workers with a Nationwide Mass Media Campaign Has Large Differential Impacts on Complementary Feeding Practices but Not on Child Growth: Results of a Cluster-Randomized Program Evaluation in Bangladesh. J Nutr. 2016 Oct;146(10):2075-2084. doi: 10.3945/jn.116.232314. Epub 2016 Aug 31. PMID 27581575